CLINICAL TRIAL: NCT01072045
Title: A Comparative Study of the Use of Beta Blocker and Oral Corticosteroid in the Treatment of Proliferative and Involuting Cutaneous Infantile Hemangioma
Brief Title: Comparative Study of the Use of Beta Blocker and Oral Corticosteroid in the Treatment of Infantile Hemangioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Dov Charles Goldenberg, Professor of Surgery, Division of Plastic Surgery, Haspital dasd Clinicas, University of Sao Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPPesq0931/09
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Hemangioma
Keywords: Hemangioma; Proliferative hemangioma; Treatment; Propranolol; Corticosteroid
MeSH Terms: conditions — Hemangioma | interventions — Propranolol; Adrenergic beta-Antagonists; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol (Active Comparator): Oral propranolol, at a dose of 2mg/kg/day, divided in 2 doses.
  Interventions: Drug: Propranolol
- Prednisone (Active Comparator): Oral prednisone , at a dose of 2mg/kg/day, divided in 2 doses.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Propranolol — Oral propranolol, at a dose of 2mg/kg/day, divided in 2 doses, for initial 60 days
  Other Names: beta-blockers
  Arms: Propranolol
Drug: Prednisone — Oral prednisone, at a dose of 2mg/kg/day, divided in 2 doses, for initial 60 days
  Other Names: corticosteroid; metilprednisolone
  Arms: Prednisone

SUMMARY:
Infantile Hemangioma (IH) is infancy's most common vascular tumor of infancy and most frequent benign neoplasm.

Treatment of IHs is indicated for approximately 10 to 20% of the cases. Two groups can be defined amongst indications for treatment: patients with absolute indication for treatment and patients with relative indication for treatment.

Absolute or emergency indications comprise function or life threatening situations such as obstruction of airways, obstruction of vision, congestive heart failure, hepatic and coagulation problems.

The following are considered relative indications: cases of large and disfiguring facial hemangiomas; locations that can result in a deformity and/ or permanent scar (nose, ear, lip, glabellar area); extensive face hemangiomas, mainly when there is dermal damage (more probable to scar); local complications such as ulceration, infection and bleeding as well as small hemangiomas in exposed areas (hands and face), mainly if pedunculated due to its ease of excision2,7.

Treatment modalities vary according to the extension, location, presence of complications and the evolutional phase. A combination of various treatments is possible.

Beta blockers are being used in children for approximately 40 years, with proven clinical safety and no cases of death or cardiovascular disease resulting from its direct use. Recently it was reported the use of beta blockers (propanolol) for IH treatment, with significant reduction of tumor volume after introduction of the beta blocker, in a short period of time, with stable results after the end of treatment, which suggested evidences of the benefits of this drug in the tumor treatment The proposal of this study is to assess the use of propanolol in IH treatment, quantifying its effectiveness and safety under continuous monitoring and comparing it to the use of oral corticosteroid. The investigators propose the assessment of the betablockers' use in comparison to the use of corticosteroids in infants with IH in the proliferative or involuting phases, with indication for clinical treatment, and that are not alarming nor urgent; in other words, the current relative indications for treatment.

DETAILED DESCRIPTION:
1. Introduction Infantile Hemangioma (IH) is infancy's most common vascular tumor of infancy and most frequent benign neoplasm. In 1996 the "International Society for the Study of Vascular Anomalies" has defined the guidelines for the diagnosis and treatment of vascular anomalies. Hemangioma is one of the many vascular tumors that were classified. Clinically, it presents well defined characteristics and a natural history divided into three phases. The proliferative phase represents an initial growth phase through hyperplasia and hypertrophy, followed by a spontaneous regression phase called the involuting phase. The involuted phase represents a final phase with no more biological activity; however, it doesn't necessarily corresponds to the complete tumor disappearance once there is a replacement by fibro-fatty tissue. IH affects one in every 10 to 20 Caucasian infants.There is a predilection for females at a 3:1 to 5:1 proportion, a higher incidence in premature infants, in newborns with low birth weight, in those whose pregnancy presented placentary anomalies and in neonates from mothers with multiple pregnancies. Fifty to sixty percent of IH affect the head and neck area.

   In the proliferative phase the tumor may reach considerable dimensions and depending on its location and proximity to vital structures, it may result in the obstruction or invasion of organs. This would cause a functional problem and even impose a threat to infant's life. There is a variable incidence of local complications such as necrosis, repetitive ulcerations, bleeding and infections, apart from systemic complications such as coagulopathy and high output cardiac failure.

   After involution, IHs may leave scars or contour deformities resulting in deformities and eventual psychological damage. Treatment of IHs is indicated for approximately 10 to 20% of the cases. Two groups can be defined amongst indications for treatment: patients with absolute indication and patients with relative indication for treatment. Absolute or emergency indications comprise function or life threatening situations such as obstruction of airways, obstruction of vision, congestive heart failure, hepatic and coagulation problems.

   The following are considered relative indications: cases of large and disfiguring facial hemangiomas; locations that can result in a deformity and/ or permanent scar (nose, ear, lip, glabellar area); extensive face hemangiomas, mainly when there is dermal damage (more probable to scar); local complications such as ulceration, infection and bleeding as well as small hemangiomas in exposed areas (hands and face), mainly if pedunculated due to its ease of excision.

   Treatment modalities vary according to the extension, location, presence of complications and the evolutional phase. A combination of various treatments is possible.

   In cases of relative indication, surgical treatment is mostly indicated for lesions in growing areas with disfiguring potential. For the other cases, pharmacological therapy is being the routine. The mostly used option is prednisone, a systemic corticosteroid administered orally. The therapeutic response to corticosteroids is variable and its effectiveness rates fluctuate between 30 to 84%. Clearly effective responses or just a reduction in the lesion's growth rate are possible. The effective response, when observed, occurs on average a week after the beginning of use of medication. Side effects are frequent, being the most common the cushingoid appearance, alterations of personality, hypertension, gastrointestinal disorders, decrease in growth speed and head circumference and weight gain.

   For cases with no response to the corticosteroid, the most frequently used drug as a second treatment line is subcutaneous alpha-interferon 2b. In spite of being very effective, this medication presents a higher rate of side effects, being spastic diplegia the most fearsome.

   Other drugs are being used, such as chemotherapeutic drugs and immunomodulators. However, published studies cover small casuistics, with no great population studies or long term follow up to justify its routine use.

   Recently, Léauté-Labrèze et al. reported the use of beta blockers (propanolol) for IH treatment. The casual finding of a significant reduction in hemangiomas volume was observed when this drug was used as an antihypertensive for the treatment of side effects resulting from the use of systemic corticoids in the treatment of infantile hemangioma. A significant reduction of tumor volume was observed after introduction of the beta blocker, in a short period of time, with stable results after the end of treatment, which suggested evidences of the benefits of this drug in the tumor treatment. Other authors also reported the successful use of the medication. Recent initial studies show the effectiveness of the isolated use of propanolol, suggesting the presence of specific action mechanisms for this medication.

   Beta blockers are being used in children for approximately 40 years, with proven clinical safety and no cases of death or cardiovascular disease resulting from its direct use. Side effects are already well established, such as bradycardia and transitory hypotension, requiring monitoring from the beginning of treatment. Besides, beta blockers reduce lipolysis, glycogenolysis and gluconeogenesis, predisposing to hypoglycaemia. It has to be used with special attention in neonates, who can present hypoglycaemia without medication.

   Beta blockers, and more precisely propanolol, appear as one more therapeutic option with apparent good results. So far in literature there are just some case reports and initial protocols about the use of this medication.

   Lesions located on the cervicofacial region with relative indication for treatment are more susceptible to visual exposure, causing discomfort to the patient and family, apart from the possibility of distortion of growing anatomical structures which will eventually evolve into deformities. The best management for these cases is debatable: on one hand the possibility of pharmacological treatment with corticosteroids with a variable success rate and significant side effects; on the other hand the conservative/ expectant treatment, in other words, waiting for evolution, expecting a complete spontaneous regression. Therefore, a drug with known reduced side effects could be a good alternative of treatment, accelerating tumor involution and allowing a quick problem solution in comparison to the expecting conduct and to the conventional pharmacological treatment.

   In this context, the proposal is to assess the use of propanolol in IH treatment, quantifying its effectiveness and safety under continuous monitoring and comparing it to the use of oral corticosteroid.

   In the present study we propose the assessment of the betablockers' use in comparison to the use of corticosteroids in infants with IH in the proliferative or involuting phases, with indication for clinical treatment, and that are not alarming nor urgent; in other words, the current relative indications for treatment.
2. Patients and Methods

Patients are going to be recruited at the Instituto de Tratamento do Câncer Infantil (Itaci) - (Infantile Cancer Treatment Institute) - ITACI - ICr-HCFMUSP and the Division of Plastic Surgery, Hospital das Clinicas, University of Sao Paulo,once eligibility, inclusion and exclusion criteria are assessed and after signature of informed consent by legally responsible parties.

2.1. Type of Study See detailed information below

2.2. Eligibility: Infants with ages up to 2 years, of both genders, carriers of clinically diagnosed infantile hemangioma in proliferative or involutive phases and relative indication for treatment.

2.3. Inclusion Criteria: see below on separate item

2.4. Exclusion Criteria: see below on separate item

2.5. Data Gathering

Once included in the study, patients are going to be subject to:

2.51. Gathering of epidemiological data concerning pregnancy, birth and family history;

2.5.2. Determination of anatomical location and dimensions of hemangioma through direct measurements and photographic study.

* Measures in centimeters on lesion's larger axis and another one perpendicular to this axis;
* Photographic measures with a measuring tape for reference on anterior and bilateral profile positions with the same photo camera and obtained by the same technician.

2.5.3. Pediatric clinical assessment of health conditions prior to the beginning of treatment, comprising the following follow-up parameters:

* Blood pressure
* Heart rate
* Oxygen Saturation
* Weight and height

2.5.4. Laboratory assessment

* glucose blood levels
* complete blood count
* assessment of renal function

2.5.5. Specific cardiac assessment

* rest electrocardiography
* echocardiography
* PA and profile thoracic radiography

2.6. Clinical Treatment Patients in Groups A and B will undergo a treatment for an initial 60-day period, unless in the presence of criteria for medication suspension (item 2.9).

The total length of the treatment is going to be determined by the effective response to the treatment. The effective response is going to be defined as a volumetric reduction of the lesion.

2.6.1 Outcome

Reduction on volume is going to be considered as effective response. It will be evaluated based on direct measurement and photographic analysis, as mentioned in item 2.5.2.

The absence of effective response after the initial 60-day period is going to be considered as treatment failure; Group A patients' medication (propanolol) is going to be suspended and Group B (prednisone) patients are going to begin a progressive dose reduction regimen until the suspension of the medication.

2.7. Follow up during treatment

During the whole period of treatment patients will be periodically evaluated as described below:

* Clinical control and lesions measure control:
* weekly in the first two months,
* twice a week in the following months.

Considering the same parameters obtained in items 2.5.2 and 2.5.3

* Monthly laboratory control until the end of treatment considering the same parameters obtained in item 2.5.4,
* Electrocardiographic examination and echocardiography at the end of the 60-day initial treatment.

2.8. Follow up after conclusion of treatment

After suspension of treatment, patients are going to maintain a periodic outpatient treatment returning after 14 days, 21 days, 1, 2 and 6 months for evaluation of clinical parameters and lesion dimensions.

Six (6) months after the conclusion of the treatment, electrocardiography, echocardiography and chest radiography are going to be repeated.

2.9. Criteria for treatment interruption:

In the event of an indication for suspension of treatment, the patient is going to be excluded from the study and is going to follow a treatment according to the group's routine indications.

2.9.1. Group A - Propranolol:

* Hypotension below percentile 90
* Bradycardia with heart rate below percentile 90
* Bronchospasm
* electrocardiographic alterations
* echocardiographic alterations
* hypoglycaemia.

2.9.2. Group B - Prednisone

- Difficult-to-control hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients with ages up to 2 years;
* Clinically diagnosed hemangioma, in proliferative or involutive phase, with relative indication for clinical treatment, as itemized:
* lesion causing alteration of regional anatomy with no systemic or functional damage and with a diameter greater than 1 centimeter, or
* lesion causing aesthetic deformity, or
* lesion causing local repetitive complications such as ulceration, bleeding or local infection, or
* lesion causing partial damage of orifices, or
* lesion causing psychological compromise.
* Absence of cardiopathy (normal physical examination, anamnesis, echocardiography, electrocardiography and thoracic radiography);
* Informed consent signed by responsible parties

Exclusion Criteria:

* Hemangioma with absolute indication for treatment, presenting a risk to function or life;
* Patients with previous treatment for infantile hemangiomas;
* Cardiac disease;
* Pulmonary disease (asthma, bronchiolitis,bronchopulmonary dysplasias)
* Raynaud syndrome;
* Pheochromocytoma;
* Altered echocardiography, even if asymptomatic

Ages: 10 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction on tumor volume, based on direct measurement (in centimeters, 2 axis) and photographic analysis (same photo camera, obtained by the same technician) | weekly in the first two months and twice a week in the following months

SECONDARY OUTCOMES:
evidence of collateral effects | weekly on the first 2 weeks and twice a week on the following months

CONTACTS AND LOCATIONS:
Overall Officials: Dov C Goldenberg, MD, Study Director — Division of Plastic Surgery - Hospital das Clinicas - University of Sao Paulo School of Medicine
Locations (1):
- Instituto de Tratamento do Câncer Infantil (Pediatric Cancer Treatment Institute) - ITACI - ICr-HCFMUSP (Instituto da Criança do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo), São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Lawley LP, Siegfried E, Todd JL. Propranolol treatment for hemangioma of infancy: risks and recommendations. Pediatr Dermatol. 2009 Sep-Oct;26(5):610-4. doi: 10.1111/j.1525-1470.2009.00975.x. PMID 19840322
- [Background] Frieden IJ, Drolet BA. Propranolol for infantile hemangiomas: promise, peril, pathogenesis. Pediatr Dermatol. 2009 Sep-Oct;26(5):642-4. doi: 10.1111/j.1525-1470.2009.00977.x. No abstract available. PMID 19840341
- [Background] Maturo S, Hartnick C. Initial experience using propranolol as the sole treatment for infantile airway hemangiomas. Int J Pediatr Otorhinolaryngol. 2010 Mar;74(3):323-5. doi: 10.1016/j.ijporl.2009.12.008. Epub 2010 Jan 13. PMID 20071038
- [Background] Buckmiller LM. Propranolol treatment for infantile hemangiomas. Curr Opin Otolaryngol Head Neck Surg. 2009 Dec;17(6):458-9. doi: 10.1097/MOO.0b013e328332a4eb. PMID 19858718
- [Background] Mousa W, Kues K, Haas E, Lauerer P, Pavlakovic H, Schon MP, Zutt M. Successful treatment of a large hemangioma with propranolol. J Dtsch Dermatol Ges. 2010 Mar;8(3):184-6. doi: 10.1111/j.1610-0387.2009.07266.x. Epub 2009 Sep 25. English, German. PMID 19788583
- [Background] Perez RS, Mora PC, Rodriguez JD, Sanchez FR, de Torres Jde L. [Treatment of infantile hemangioma with propranolol]. An Pediatr (Barc). 2010 Feb;72(2):152-4. doi: 10.1016/j.anpedi.2009.05.019. Epub 2009 Jul 23. No abstract available. Spanish. PMID 19631595
- [Background] Denoyelle F, Leboulanger N, Enjolras O, Harris R, Roger G, Garabedian EN. Role of Propranolol in the therapeutic strategy of infantile laryngotracheal hemangioma. Int J Pediatr Otorhinolaryngol. 2009 Aug;73(8):1168-72. doi: 10.1016/j.ijporl.2009.04.025. Epub 2009 May 29. PMID 19481268
- [Background] Michel JL, Patural H. [Response to oral propranolol therapy for ulcerated hemangiomas in infancy]. Arch Pediatr. 2009 Dec;16(12):1565-8. doi: 10.1016/j.arcped.2009.09.008. Epub 2009 Nov 4. French. PMID 19892536
- [Background] Siegfried EC, Keenan WJ, Al-Jureidini S. More on propranolol for hemangiomas of infancy. N Engl J Med. 2008 Dec 25;359(26):2846; author reply 2846-7. doi: 10.1056/NEJMc086443. No abstract available. PMID 19109584
- [Background] Leaute-Labreze C, Taieb A. [Efficacy of beta-blockers in infantile capillary haemangiomas: the physiopathological significance and therapeutic consequences]. Ann Dermatol Venereol. 2008 Dec;135(12):860-2. doi: 10.1016/j.annder.2008.10.006. Epub 2008 Nov 20. No abstract available. French. PMID 19084699
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- See also: website of the International Society for the Study of Vascular Anomalies — http://www.issva.org